CLINICAL TRIAL: NCT06080646
Title: Reward Processing and Depressive Subtypes: Identifying Neural Biotypes Related to Suicide Risk, Resilience, and Treatment Response
Brief Title: Reward Processing and Depressive Subtypes: Identifying Neural Biotypes
Status: Recruiting | Type: Observational
Sponsor: San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, Susanna Fryer, PhD, Staff Psychologist/Clinician Investigator, San Francisco Veterans Affairs Medical Center
Other Study IDs: CX001980
Record Dates: First submitted 2023-09-28; First posted 2023-10-12 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Depression; Depressive Disorder; Major Depressive Disorder; Major Depressive Episode; Depressive Symptoms; Anhedonia
Keywords: reward; motivation; EEG; fMRI; MRI; functional MRI; amotivation; avolition; suicidality; suicide
MeSH Terms: conditions — Depression; Depressive Disorder; Depressive Disorder, Major; Anhedonia; Suicidal Ideation; Suicide

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MDD (Major Depressive Disorder) Group: Individuals (ages 18-70 years) who meet DSM-5 criteria for MDD, as assessed using the Structured Clinical Interview for DSM-5 (SCID-5), with Stable psychiatric medication regime for > 1 month will be recruited for participation in EEG and fMRI sessions in this observational study.
  Interventions: Other: cross-sectional MRI and EEG assessments (NO INTERVENTION)
- Unaffected Comparison Group: 50 unaffected comparison participants will be matched as a group to the age, race, educational level, handedness, and parental socio-economic status of the MDD patient group will be recruited for participation in EEG and fMRI testing sessions identical to those administered to the patients
  Interventions: Other: cross-sectional MRI and EEG assessments (NO INTERVENTION)

INTERVENTIONS:
Other: cross-sectional MRI and EEG assessments (NO INTERVENTION) — n/a there is no intervention in this observational study
  Other Names: cross-sectional MRI and EEG assessments

SUMMARY:
Deficits in motivation and pleasure are common in depression, and thought to be caused by alterations in the ways in which the brain anticipates, evaluates, and adaptively uses reward-related information. However, reward processing is a complex, multi-circuit phenomenon, and the precise neural mechanisms that contribute to the absence or reduction of pleasure and motivation are not well understood. Variation in the clinical presentation of depression has long been a rule rather than an exception, including individual variation in symptoms, severity, and treatment response. This heterogeneity complicates understanding of depression and thwarts progress toward disease classification and treatment planning. Discovery of depression-specific biomarkers that account for neurobiological variation that presumably underlies distinct clinical manifestations is critical to this larger effort.

DETAILED DESCRIPTION:
This study combines clinically motivated questions with in-depth study of neurobiological mechanisms to evaluate how reward system neurobiology contributes to expression of reward-related deficits, such as decreased pleasure and motivation in major depressive disorder (MDD). Conceptually, the investigator will use a multi-measure approach, by studying basic brain responses to reward anticipation as well as higher-order aspects of reward processing necessary for decision-making.

Methodologically, the investigator will combine fMRI, EEG, and behavioral assessment, to more fully characterize reward-related brain functions and their clinical correlates. In addition to evaluating reward effects between MDD and healthy controls (HC), the investigator will also focus on understanding the relationship between reward processing and clinical features of high relevance to depression, with an emphasis on suicidality.

ELIGIBILITY:
* Our studies require some in-person visits to our research lab, located at 42nd Ave and Clement St in San Francisco.
* Because this study includes an MRI, part of the screening process will be to ensure you don't have any metal in your body, you do not have head or neck tattoos, and you are comfortable inside the MRI scanner.

Inclusion Criteria:

* 18-70 years with a diagnosis of major depressive disorder (MDD) for MDD group, or without for unaffected comparison (UC) group
* Negative metal screen for MRI safety
* Normal (or corrected to normal) vision

Exclusion Criteria:

* Past or present neurological problems (including seizures and head trauma resulting in neurological or cognitive symptoms)
* Loss of consciousness (LOC) greater than 30 minutes or any LOC with neurologic symptoms
* Major medical conditions (e.g., seizure disorders, treatment with anticonvulsant medication, endocrine disorders, significant cardiac pathology)
* Substance dependence, within the past year, or failed urine toxicology on the day of neuroimaging sessions
* Known claustrophobia
* Current Pregnancy
* IQ estimate < 70

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals with Major Depressive Disorder (age range 18 - 70)
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Stimulus preceding negativity | 1 month (EEG measure of reward anticipation)
  Stimulus preceding negativity (EEG measure of reward anticipation) of reward-related brain activation patterns and EEG responses on participants
Reward positivity | 1 month (EEG measure of reward feedback)
  Reward positivity (EEG measure of reward feedback) of reward-related brain activation patterns and EEG responses on participants
Late positive potential | 1 month (EEG measure of effective salience)
  Late positive potential (EEG measure of affective salience) of reward-related brain activation patterns and EEG responses on participants
fMRI response to win vs. loss reward feedback | 1 month (fMRI data)
  fMRI response to win vs. loss reward feedback of reward-related brain activation patterns and EEG responses on participants

CONTACTS AND LOCATIONS:
Overall Officials: Susanna L Fryer, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- San Francisco Healthcare System, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No
Not part of currently approved protocol or original agreement with sponsor